CLINICAL TRIAL: NCT03672968
Title: EAP Single Patient: Safety of Bilateral Intravitreal Injection of GS010 in a Single Subject Affected With G11778A ND4 Leber Hereditary Optic Neuropathy
Brief Title: EAP_GS010_single Patient
Status: No longer available | Type: Expanded Access
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP_GS010_001
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Leber Hereditary Optic Neuropathy (Optic, Atrophy, Hereditary, Leber)
Keywords: Heredity Optic Atrophy; Leber Hereditary Optic Atrophy; Leber Hereditary Optic Neuropathy; LHON; Eye Diseases; Hereditary Eye Diseases; Inherited retinal dystrophies or degeneration; Inborn Genetic Disease; Gene Therapy; Intravitreal Injections; Mitochondrial Disease; AAV2 Vectors; Neurodegenerative Disease; Atrophy
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Atrophy; Eye Diseases; Eye Diseases, Hereditary; Genetic Diseases, Inborn; Mitochondrial Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Genetic: GS010

SUMMARY:
Expanded Access Use for a single patient of Bilateral Intravitreal Injection of GS010 in a Single Subject Affected with G11778A ND4 Leber Hereditary Optic Neuropathy

ELIGIBILITY:
The EAP applies to patients not eligible to ongoing GS010 clinical trials.

Inclusion Criteria:

* Presence of documented G11778A ND4 LHON-causing mutation
* Signature of informed consent and assent from the parent/guardian and the patient.

Exclusion Criteria:

Contraindications to GS010 product or IVT procedures are to be checked prior to consent signature and treatment injection:

* Any known allergy or hypersensitivity to GS010 or its constituents.
* Contraindication to intravitreal injection in any eye.
* Intravitreal drug delivery to any eye within 30 days prior to the injection
* Previous vitrectomy in either eye.
* Narrow angle in any eye contra-indicating pupillary dilation.
* Presence of disorders or diseases of the eye or adnexa, excluding LHON, which may interfere with visual or ocular assessments, including SD-OCT, during the study period.
* Presence of known/documented mutations, other than the G11778A ND4 LHON-causing mutation, which are known to cause pathology of the optic nerve, retina or afferent visual system.
* Presence of systemic or ocular/vision diseases, disorders or pathologies, other than LHON, known to cause or be associated with vision loss, or whose associated treatment(s) or therapy(ies) is/are known to cause or be associated with vision loss.
* Presence of optic neuropathy from any cause except LHON.
* Presence of illness or disease that, in the opinion of the Investigator, include symptoms and/or the associated treatments that can alter visual function, for instance cancers or pathology of the central nervous system, including Multiple Sclerosis (diagnosis of Multiple Sclerosis must be based on the 2010 Revisions to the McDonald Criteria [Polman 2011]).
* History of recurrent uveitis (idiopathic or immune-related) or active ocular inflammation.
* Previous treatment with ocular gene therapy in either eye.
* Subjects who have undergone ocular surgery of clinical relevance (per Investigator assessment) within 90 days prior to injection.
* Subjects who are unable to tolerate (e.g. the immune modulating regimen) or unable or unwilling to comply with all the protocol requirements.

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Related Info — http://www.gensight-biologics.com